CLINICAL TRIAL: NCT01200329
Title: High-Dose Gemcitabine, Busulfan and Melphalan With Hematopoietic Cell Support for Patients With Relapsed/Refractory Hodgkin's Disease
Brief Title: High-Dose Gemcitabine, Busulfan and Melphalan for Patients With Refactory Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0142; NCI-2012-01885 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Lymphoma
Keywords: Hodgkin's disease; Relapsed; Refractory; High-dose chemotherapy; Busulfan; Gemcitabine; Melphalan
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence | interventions — Gemcitabine; Busulfan; Melphalan; Stem Cell Transplantation; Fibroblast Growth Factor 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcitabine + Busulfan + Melphalan (Experimental): Gemcitabine 2775 mg/m2 by vein over about 3 hours on days -8 and -3. Busulfan 32 mg/m2 test dose with PKs as outpatient and on day -10 as inpatient. AUC 4,000 by vein over about 3 hours on days -8 to -5. Melphalan 60 mg/m2 by vein over about 30 minutes on days -3 and -2. Palifermin 60 mg/kg by vein over 30 seconds daily, Days -12 to -10 and Days 0 to 2. Infusion of stem cells on Day 0.
  Interventions: Drug: Gemcitabine; Drug: Busulfan; Drug: Melphalan; Procedure: Stem Cell Transplantation; Drug: Palifermin

INTERVENTIONS:
Drug: Gemcitabine — 2775 mg/m2 by vein over about 3 hours on days -8 and -3.
  Other Names: Gemcitabine Hydrochloride; Gemzar
Drug: Busulfan — 32 mg/m2 test dose with PKs as outpatient and on day -10 as inpatient
  AUC 4,000 by vein over about 3 hours on days -8 to -5.
  Other Names: Busulfex; Myleran
Drug: Melphalan — 60 mg/m2 by vein over about 30 minutes on days -3 and -2.
  Other Names: Alkeran
Procedure: Stem Cell Transplantation — Infusion of stem cells on Day 0.
  Other Names: SCT
Drug: Palifermin — 60 mg/kg by vein over 30 seconds daily, Days -12 to -10 and Days 0 to 2.
  Other Names: Kepivance

SUMMARY:
The goal of this clinical research study is to learn if the combination of gemcitabine, busulfan, and melphalan, when given before a stem cell transplant, can help to control refractory Hodgkin's disease. The safety of this study treatment will also be studied.

DETAILED DESCRIPTION:
Study Drugs:

Busulfan and melphalan are designed to kill cancer cells by binding to DNA (the genetic material of cells), which may cause cancer cells to die. They are commonly used in stem cell transplantation.

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause cancer cells to die. It may help to increase the effect of busulfan and melphalan on cancer cells by not allowing these cells to repair the DNA damage caused by busulfan or melphalan.

Apheresis:

Your cells have previously been collected by a procedure called apheresis. Apheresis is the process of filtering part of the blood from the body in order to remove the stem cells. The rest of the blood is then returned back to your body. You signed a separate consent for this procedure.

Busulfan Test Dose:

You will receive a test dose of busulfan by vein over about 1 hour. This low-level test dose of busulfan is to check how the level of busulfan in your blood levels changes over time. This information will be used to decide the next dose needed to reach the target blood level that matches your body size. You will most likely receive this as an outpatient during the week before you are admitted to the hospital. If it cannot be given as an outpatient, you will be admitted to the hospital on Day -11 (11 days before your stem cells are returned to your body) and the test dose will be given on Day -10.

About 11 samples of blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing of busulfan. PK testing measures the amount of study drug in the body at different time points and will help the study doctor determine what your dose of busulfan should be on study. These blood samples will be drawn at various timepoints before you receive busulfan and over about the next 11 hours. The blood samples will be repeated again on the first day of high-dose busulfan treatment (Day -8). A temporary heparin lock line will be placed in your vein to lower the number of needle sticks needed for these draws. If it is not possible for the PK tests to be performed for technical or scheduling reasons, you will receive the standard fixed dose of busulfan.

If you receive the busulfan test dose as an outpatient:

On Days -12 through Day -10, you will receive palifermin by vein over about 30 seconds each day to help decrease the risk of side effects in the mouth and throat.

You will be admitted on Day -9 and will receive fluids by vein. You will begin to swish the liquids caphosol and glutamine in your mouth 4 times a day, for about 2 minutes each time. You will swish these liquids every day until you leave the hospital. These drugs are also used to help decrease the risk of side effects in the mouth and throat.

If you receive the busulfan test dose as an inpatient:

On Days -13 through Day -11, you will receive palifermin by vein over about 30 seconds each day to help decrease the risk of side effects in the mouth and throat.

You will be admitted on Day -11 and will receive fluids by vein. You will begin to swish the liquids caphosol and glutamine in your mouth 4 times a day, for about 2 minutes each time. You will swish these liquids every day until you leave the hospital. These drugs are also used to help decrease the risk of side effects in the mouth and throat.

On Day -10 you will receive the Busulfan test dose by vein over 1 hour.

Study Drug Administration (for all patients):

On Days -9 through -2, you will receive dexamethasone by vein over about 15 minutes to help decrease the risk of the possible side effects of the study drugs.

On Days -8 through -5, you will receive busulfan by vein over about 3 hours each day.

On Days -8 and -3, you will receive gemcitabine by vein over about 4 hours on both days.

On Days -3 and -2, you will receive melphalan by vein over about 30 minutes on both days.

On Day -1, you will not receive any study drugs.

On Day 0, your stem cells will be returned to your body by vein over 30-60 minutes.

On Days 0 through 2, you will receive palifermin by vein over about 30 seconds each day.

Beginning on Day +5, you will receive filgrastim (a drug that helps with the growth of white blood cells) through a needle under your skin 1 time each day until your blood cell levels return to normal.

If your tumor cells are found to have the CD20 protein, you will receive rituximab by vein over 4-8 hours on Days 1 and 8, which is standard treatment for this type of tumor when combined with high-dose chemotherapy.

Study Tests:

While you are in the hospital, you will be checked for any side effects as part of your standard of care. Blood (about 2 teaspoons) will be drawn every day to check for side effects.

As part of standard care, you will remain in the hospital for about 3-4 weeks after transplantation. After you are released from the hospital, you must remain in the Houston area to be monitored for infections and other transplant side effects until about Day 30. During this time, you will return to the clinic 1 time each week and the following tests and procedures will be performed:

* You will be asked about how you are feeling and about any side effects you may be having.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Around Day 30, if your doctor thinks it is needed, you will have a positron-emission tomography/CT (PET/CT) and/or a CT scan of the chest, abdomen, and pelvis to check the status of the disease.

You will have a lung function test about 30-100 days after the transplant.

Length of Study:

You will be taken off study about 100 days after the transplant. You may be taken off study early if the disease gets worse or you experience any intolerable side effects.

You must talk to the study doctor if you want to leave the study early. It may be life-threatening to leave the study after you have begun to receive the study drugs but before you receive the stem cells.

End-of-Study Visit:

At Day 100, the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a physical exam.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* If your doctor thinks it is needed, you will have a (PET/CT) and/or a CT scan of the chest, abdomen, and pelvis to check the status of the disease.
* If your doctor thinks it is needed, you will have a bone marrow biopsy to check the status of the disease.

This is an investigational study. Busulfan, gemcitabine, and melphalan are all FDA approved and commercially available for the treatment of lymphoma and several other tumors. The use of these study drugs together and the use of gemcitabine at the dose level used in this study is investigational.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 to 70 years
2. Patients with relapsed Hodgkin's disease and one or more of the following: 1) Less than complete response to first-line chemotherapy, 2) Relapse within 12 months of completion of first-line chemotherapy, 3) Relapse within a prior irradiation field, 4) Less than complete metabolic response to second-line chemotherapy, 5) Second relapse or beyond, 6) Extranodal disease at the time of relapse, 7) Presence of B symptoms at the time of persistent disease upon completion of first-line chemotherapy, or of relapse, progressive disease, 8) Bulky disease (defined as any lesion greater than 5 cm) at the time of persistent disease upon completion of first-line chemotherapy, or of relapse, progressive disease.
3. Adequate renal function, as defined by estimated serum creatinine clearance >/=50 ml/min (using the Cockcroft-Gault formula: creatinine clearance = [(140-age)*kg/(72*serum creatinine)] * 0.85 if female) and/or serum creatinine </=1.8 mg/dL.
4. Adequate hepatic function, as defined by SGOT and/or SGPT </=3 x upper limit of normal; serum bilirubin and alkaline phosphatase </=2 x upper limit of normal, unless due to disease involvement
5. Adequate pulmonary function with FEV1, FVC and DLCO >/=50% of expected corrected for hemoglobin and/or volume.
6. Adequate cardiac function with left ventricular ejection fraction >/=40%. No uncontrolled arrhythmias or symptomatic cardiac disease.
7. Zubrod performance status <2.
8. Negative Beta HCG text in a woman with child-bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization

Exclusion Criteria:

1. Patients with grade >/= 3 non-hematologic toxicity from previous therapy that has not resolved to </= grade 1.
2. Patients with prior whole brain irradiation
3. Patients with active hepatitis B, either active carrier (HBsAg +) or viremic (HBV DNA >/=10,000 copies/mL, or >/= 2,000 IU/mL).
4. Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology.
5. Active infection requiring parenteral antibiotics.
6. HIV infection, unless the patient is receiving effective antiretroviral therapy with undetectable viral load and normal CD4 counts
7. Patients having received radiation therapy to head and neck (excluding eyes), and internal organs of chest, abdomen or pelvis in the month prior to enrollment.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yago Nieto, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Nieto Y, Gruschkus S, Valdez BC, Jones RB, Anderlini P, Hosing C, Popat U, Qazilbash M, Kebriaei P, Alousi A, Saini N, Srour S, Rezvani K, Ramdial J, Barnett M, Gulbis A, Shigle TL, Ahmed S, Iyer S, Lee H, Nair R, Parmar S, Steiner R, Dabaja B, Pinnix C, Gunther J, Cuglievan B, Mahadeo K, Khazal S, Chuang H, Champlin R, Shpall EJ, Andersson BS. Improved outcomes of high-risk relapsed Hodgkin lymphoma patients after high-dose chemotherapy: a 15-year analysis. Haematologica. 2022 Apr 1;107(4):899-908. doi: 10.3324/haematol.2021.278311. PMID 33951890
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled at MD Anderson clinic starting on June 16, 2011.
Groups:
- Overall Study Group: Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto Stem Cell Transplant (SCT)+Palifermin 60 mcg/kg IV for 3 days post SCT
Period: Overall Study
Arm/Group | Overall Study Group
Started | 81
Completed | 78
Not Completed | 3
Not completed — Lack of financial coverage | 2
Not completed — Progressive disease | 1

BASELINE CHARACTERISTICS:
Population: Patients with relapsed/refractory Hodgkin's disease (ie, extranodal relapse or within 1 year of frontline therapy).
Arm/Group | Overall Study Group
Number analyzed (Participants) | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 74
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 31.5 [13 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 52
  More than one race | 0
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  United States | 78
Overall Study Group [Number; unit: participants] — For patients with primary refractory Hodgkin's, they either progressed or had no response to front-line therapy. For patients with relapsed Hodgkin's, they relapsed within the 1st year to front-line therapy or had extranodal relapse.
  participants
    Primary Refractory Hodgkin's | 32
    Relapsed Hodgkin's | 46

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) of Patients
Description: The event-free survival (EFS) of patients with poor prognosis relapse or refractory Hodgkin's disease (HD) after high-dose chemotherapy (HDC) with Gemcitabine/Busulfan/Melphalan (GemBuMel). Event is defined as relapse, tumor progression or death.Progression free survival is the length of time during and after the treatment of disease that a patient lives with the disease but it does not get worse. Toxicity is defined as the treatment related mortality (TRM) rate, which will be evaluated within 30 days post transplant, and this rate will be compared with the 5% maximum rate. For EFS analysis, patients who experience the tumor relapse, disease progression, or death will be considered to be an event.
Time Frame: Enrollment up to 2 years post transplant
Population: Patients with relapsed/refractory Hodgkin's disease (ie, extranodal relapse or within 1 year of frontline therapy).
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 78
Participants | 51

2. Secondary Outcome: Overall Survival (OS) of These Patients.
Description: The overall survival is the length of time from the start of treatment (Auto SCT) for the cancer, that patients are diagnosed with are still alive until date of first documented progression or date of death from any cause. It is measured in months and assessed up to 84 months.
Time Frame: Beyond 100 days post transplant up to 84 months.
Measure: Median (Full Range); unit: Months
Arm/Group | Overall Study Group
Number analyzed (Participants) | 78
Months | 52 [4 to 84]

ADVERSE EVENTS:
Time Frame: Up to 100 Days post transplant
Arm/Group | Overall Study Group
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 78/78
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study Group (N=78)
Hypertension (Cardiac disorders) | 5 (5)
Fluid Overload (General disorders) | 33 (33)
Fever (General disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 39 (40)
Mucositis (Gastrointestinal disorders) | 76 (76)
Nausea (Gastrointestinal disorders) | 68 (68)
Transaminitis (Hepatobiliary disorders) | 55 (63)
Elevated Bilirubin (Hepatobiliary disorders) | 36 (36)
Infection (Infections and infestations) | 20 (27)
Neutropenic Fever (General disorders) | 62 (62)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Skin Rash (Skin and subcutaneous tissue disorders) | 53 (54)
Skin Hand/Foot Syndrome (Skin and subcutaneous tissue disorders) | 6 (6)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4)
Headache (Nervous system disorders) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT01200329/Prot_SAP_000.pdf